CLINICAL TRIAL: NCT01103388
Title: Maintenance Therapy With Rituximab After Autologous Transplantation for Non-Hodgkin's Lymphoma
Brief Title: Rituximab Maintenance After Autologous Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed early due to slow patient accrual and sponsor's withdrawal of support.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0239
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Rituximab; Rituxan; Lymphoma; High dose chemotherapy; Autologous transplantation; Autologous stem cell transplant; ASCT
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab
- No Rituximbab (No Intervention)

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2 by vein (IV) in 4 weekly doses (1 cycle) every 6 months for 4 cycles.
  Other Names: Rituxan
  Arms: Rituximab

SUMMARY:
The goal of this clinical research is to see if Rituxan (rituximab) therapy given after high dose chemotherapy and transplant of a patients own stem cells will prevent or delay the return of the lymphoma.

DETAILED DESCRIPTION:
Rituxan is a mouse antibody that has been changed to make it similar to a human antibody. Antibodies are proteins that can protect the body from foreign invaders, such as bacteria and viruses, by binding to substances called antigens. Rituxan works by binding to a protein, called the CD20 protein (which is found on the surface of normal and cancerous B-lymphocytes). This binding may help to destroy the B-lymphocytes.

Before the study begins, you will have a physical exam, routine blood tests (1-2 tablespoons), and urine tests. Women who are able to have children must have a negative blood pregnancy test. You will also have a chest x-ray and an ECG (test to measure the electrical activity of the heart). The status of the lymphoma will be evaluated by bone marrow biopsy. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. CT scans and gallium or PET scans will be performed. If you had lymphoma in other areas of your body additional tests may be needed as determined by your treating physician. Tests to evaluate the status of the lymphoma will be repeated before each cycle of chemotherapy. If your white count is low you may need injections of NeupogenTM (growth factor) daily till your white blood cell count is high enough to start the next round of treatment.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive rituximab. Participants in the other group will not receive rituximab. There is an equal chance of being assigned to either group.

Treatment will start between 5-6 months after your stem cell transplant. If you are assigned to the rituximab group, you will receive a total of 4 cycles of treatment. Each cycle will be given 6 months apart. Each cycle is made up of 4 doses of rituximab given once a week for 4 weeks. If the disease returns or intolerable side effects occur while on treatment, you will be taken off the study. You may still be able to receive rituximab outside of this study if your treating physician decided that it is okay.

Treatment will be given on an outpatient basis. The treatment can be given at M. D. Anderson or by your local cancer doctor. Patients who are assigned to the rituximab arm must be willing to get their first and third cycle (all 4 doses) at M. D. Anderson, if their local physician is unable to draw and ship samples to the central laboratory for rituximab levels. Blood will be drawn (approximately one teaspoon) before and after the first and fourth dose and before the second and third dose of those two treatment cycles. The treatment will be given by vein over a period of several hours. Participants who have easily accessible veins may get this treatment by having a temporary needle placed in the vein for the treatment. For participants who do not have easily accessible veins, a central venous catheter (long plastic tube - CVL) will be placed in a big vein of the arm or chest.

Participants who do not receive rituximab will be followed every 6 months at M. D. Anderson as is standard of care.

All participants (even those who do not receive the rituximab) will have to return to M. D. Anderson every 6 months for a period of 3 years (from the date of enrollment) to have the lymphoma evaluated. The status of the lymphoma will be evaluated by blood tests (1-2 tablespoons), CT scans, PET or Gallium scans and bone marrow biopsy.

This is an investigational study. Rituximab has been approved by the FDA. About 90 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diffuse large B cell non-Hodgkin's lymphoma who are 5-6 months status post an autologous stem cell transplant and are in CR. Patients who are positive for t(14;18) by PCR or for BCL-2 by Southern blot are eligible provided there is no other disease present.
2. Absolute neutrophil count (ANC) > 1500/mm3 independent of growth factor support
3. No evidence of symptomatic cardiac or pulmonary disease
4. Platelet count > 75,000 mm3
5. Zubrod performance status of 2 or less.
6. Negative pregnancy test in patients of "child bearing potential"

Exclusion Criteria:

1. Uncontrolled active infection
2. Severe concomitant medical or psychiatric illness
3. Serum bilirubin > 2.0 mg/dl 4) Transaminases > 2xULN 5) Serum creatinine > 2.0 mg/dl

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-08; Primary Completion 2006-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Progression Free Survival (PFS) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org